CLINICAL TRIAL: NCT01967758
Title: Phase I Study of Safety and Immunogenicity of ADU-623, a Live-attenuated Listeria Monocytogenes Strain (ΔactA/ΔinlB) Expressing the EGFRvIII-NY-ESO-1 Vaccine, in Patients With Treated and Recurrent WHO Grade III/IV Astrocytomas
Brief Title: Phase I Study of Safety and Immunogenicity of ADU-623
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Providence Health & Services (Other)
Collaborators: Aduro Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-012A
Record Dates: First submitted 2013-10-18; First posted 2013-10-23 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Astrocytic Tumors; Glioblastoma Multiforme; Anaplastic Astrocytoma; Brain Tumor
Keywords: Astrocytic Tumors; Glioblastoma Multiforme; Anaplastic Astrocytoma; Brain Tumor; Brain Cancer; Immunotherapy
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Brain Neoplasms | interventions — KPNA1 protein, human; Anti-Bacterial Agents; Amoxicillin; Amoxicillin-Potassium Clavulanate Combination; Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Experimental): Patients in Cohort 1 will receive ADU-623 at a dose of 3 x 10^7cfu by intravenous infusion (IV) over 2 hours on Day 0, Day 21, Day 42, and Day 63. Each dose is followed by a 3-day course or antibiotics. Patients will receive a 7-day course of antibiotics starting at the end of treatment visit.
  Interventions: Biological: Cohort 1; Drug: Antibiotics
- Cohort 2 (Experimental): Patients in Cohort 2 will receive ADU-623 at a dose of 3 x 10^8cfu by intravenous infusion (IV) over 2 hours on Day 0, Day 21, Day 42, and Day 63. Each dose is followed by a 3-day course or antibiotics. Patients will receive a 7-day course of antibiotics starting at the end of treatment visit.
  Interventions: Biological: Cohort 2; Drug: Antibiotics
- Cohort 3 (Experimental): Patients in Cohort 3 will receive ADU-623 at a dose of 3 x 10^9cfu by intravenous infusion (IV) over 2 hours on Day 0, Day 21, Day 42, and Day 63. Each dose is followed by a 3-day course or antibiotics. Patients will receive a 7-day course of antibiotics starting at the end of treatment visit.
  Interventions: Biological: Cohort 3; Drug: Antibiotics

INTERVENTIONS:
Biological: Cohort 1 — Four doses of IV ADU-623 at a dose of 3 x 10^7cfu
  Arms: Cohort 1
Biological: Cohort 2 — Four doses of IV ADU-623 at a dose of 3 x 10^8cfu
  Arms: Cohort 2
Biological: Cohort 3 — Four doses of IV ADU-623 at a dose of 3 x 10^9cfu
  Arms: Cohort 3
Drug: Antibiotics — A 3-day course of oral amoxicillin (500 mg three times per day) or trimethoprim/sulfamethoxazole in penicillin-allergic patients (160 mg trimethoprim / 800mg sulfamethoxazole at 12 hour intervals) will be initiated for each patient 3 days following each dose of ADU-623. Patients will receive a 7-day course of antibiotics starting at the end of treatment visit.
  Other Names: Amoxicillin; Augmentin; trimethoprim / sulfamethoxazole; Bactrim

SUMMARY:
This is a study for patients with brain tumors called astrocytic tumors. The study will enroll patients who have received standard treatment. The study will test a vaccine called ADU-623. ADU-623 has not been tested in humans before, so the goal of this study is to see if ADU-623 can be given safely to brain cancer patients and what is the better dose to give patients among the three doses that planned to be tested. This study will also evaluate the length of time before patients' cancer worsens and if ADU-623 helps patients to live longer. The study will also measure the body's immune system response to ADU-623.

DETAILED DESCRIPTION:
This Phase I clinical trial will examine the safety, tolerability and immunogenicity of a novel vaccine approach using a live-attenuated strain of Listeria monocytogenes expressing EGFRvIII and NY-ESO-1 antigens to induce proliferation of memory and effector T cells with the overall goal of promoting an immune response against high-grade astrocytic tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a pathologic diagnosis of WHO Grade III or Grade IV astrocytic tumors that have completed standard of care or with radiographic evidence of progression following standard of care.
* Tumor tissue blocks available to perform both EGFRvIII and NY-ESO-1 testing
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 or Karnofsky Performance Status (KPS) 70-100
* Age 18 years or above
* Have a life expectancy of more than 12 weeks
* Laboratory values (performed within 5 days) within designated range.
* For women and men of childbearing potential, an acceptable method of highly effective contraception
* Ability to give informed consent and comply with the protocol.

Exclusion Criteria:

* Have a known allergy to both penicillin and sulfa
* Have artificial (prosthetic) joint(s), orthopedic screw(s), metal plate(s) or other exogenous implant(s) or device(s) that cannot be easily removed (i.e., prosthetic heart valves).
* Have any evidence of hepatic cirrhosis or clinical or radiographic ascites.
* Have radiographic or clinically significant pleural effusion.
* Receipt of prophylactic vaccine within 28 days of study treatment.
* Unable to avoid close contact with another individual known to be at high risk of listeriosis (e.g., newborn infant, pregnant woman, HIV-positive individual).
* History of allergy to yeast or any other component of the ADU-623 vaccine (e.g., glycerol).
* Have an immunodeficiency disease or immunocompromised state (e.g., use of immunosuppressive agents; chemotherapy or radiation therapy within 14 days of study treatment).
* Have had major surgery or significant traumatic injury occurring within 28 days before treatment administration or anticipated surgery or procedure requiring general anesthesia during study participation (including 28 days after last dose of ADU-623).
* Use of more than 4 grams per day of acetaminophen.
* Have received an investigational product within 28 days of study treatment or planned to receive within 28 days after vaccine administration.
* Have an unhealed surgical wound.
* Have clinically significant heart disease (such as uncontrolled angina, myocardial infarction with the last 3 months, congestive heart failure of New York Heart Association III or IV).
* Have valvular heart disease that requires antibiotic prophylaxis for prevention of endocarditis.
* Have an intercurrent illness that is either life-threatening or of clinical significance such that it might limit compliance with study requirements including, but not limited to, ongoing or active infection, metabolic or neurological disease, peripheral vascular disease or psychiatric illness.
* Have insufficient peripheral venous access to permit completion of the study dosing and compliance with study phlebotomy regimen.
* Have received a diagnosis of HIV, HCV, or HBV (patients with hepatitis C antibody positive may be enrolled if they are confirmed with negative viral load at screening).
* Have an active autoimmune disease or history of autoimmune disease requiring systemic steroids or other immunosuppressive treatment.
* Other medical or psychiatric conditions that in the opinion of the Principal Investigator would preclude safe participation in protocol.
* Pregnant or lactating women, as treatment has unknown effect on the embryo or child.
* Patients requiring chronic corticosteroid use will be excluded as this may mask toxic effects related to the vaccine and may prevent the development of effective immune responses following vaccination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-01-08 (Actual); Primary Completion 2018-06-18 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 91 Days
  The primary objective of this trial is to determine the maximum tolerated dose (MTD)(up to a dose of 1x10^9 cfu IV) and characterize the safety profile of ADU-623 vaccine in patients with recurrent WHO Grade III/IV Astrocytomas. The MTD will be defined as the highest dose at which none or one out of 6 patients experiences a dose-limiting toxicity (DLT) that is possibly or probably related to the vaccine.

SECONDARY OUTCOMES:
Tumor response based on magnetic resonance imaging (MRI) exam | 24 months
  The efficacy of therapy on tumor burden and time to progression will be assessed by MRI.
Immune Response | 91 Days
  Innate and adaptive immunologic response will be assessed by looking at changes in cytokines and changes in cellular and humoral immunity.

CONTACTS AND LOCATIONS:
Overall Officials: Marka Crittenden, MD, PhD, Principal Investigator — Providence Health & Services
Locations (1):
- Providence Cancer Center, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
Data generated by this study will be shared with the collaborator, Aduro BioTech.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data has been available from study start-up through the end of data analysis. Anticipated August 2018.
Access Criteria: De-identified data will be made available to Aduro BioTech.

REFERENCES:
- See also: Providence Cancer Center — https://oregon.providence.org/our-services/p/providence-cancer-center/